CLINICAL TRIAL: NCT06749665
Title: Efficacy and Safety of Intralesional Injections of Candida Antigen, Polidocanol Sclerotherapy and Combined Candida Antigen With Polidocanol in Treatment of Patients With Common Warts
Brief Title: Sclerotherapy and Candida Antigen in Treatment of Common Warts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Heba Shawky Osman, Resident at Dermatology, Venereology, and Andrology Department Sohag University Hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HShawkyosman
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Common Wart
MeSH Terms: conditions — Warts | interventions — PRA1 protein, Candida albicans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Polidacanol (Active Comparator): will receive intralesional injection of (polidacanol 3% (Aethoxysklerol 3%,60mg/ ml ampoule, kreussler pharma, Germany) During the study, the dosage of the drug and frequency of treatment will be uniform in all patients. The base of each wart will inject until the lesion blanch using an insulin syringe (29 Gage × 0.5-in) every 2 weeks until the resolution of warts or for a maximum of 6 sessions.
  Interventions: Drug: polidacanol 3%
- Candida (Active Comparator): will receive intralesional injection of candida antigen at a dose of 0.2 ml. Each treatment will inject into the largest wart using an insulin syringe (29 Gage × 0.5-in) every 2 weeks until complete clearance of warts or for a maximum of 6 treatment sessions.
  Interventions: Biological: candida antigen
- Polidacanol and candida (Active Comparator): will receive intralesional candida antigen injection in the largest wart and intralesional injection of (polidacanol 3%) in all warts using an insulin syringe (29 Gage × 0.5-in) every 2 weeks until complete clearance of warts or for a maximum of 6 treatment sessions
  Interventions: Drug: polidacanol 3%; Biological: candida antigen

INTERVENTIONS:
Drug: polidacanol 3% — Aethoxysklerol 3%,60mg/ ml ampoule, kreussler pharma, Germany
  Arms: Polidacanol; Polidacanol and candida
Biological: candida antigen — delayed type of hypersensitivity reaction is induced toward the injected antigen and the wart virus as well. This can increase the ability of the immune system to recognize and eradicate the human papillomavirus on various parts of the body and eliminate the necessity of local treatment for each wart
  Arms: Candida; Polidacanol and candida

SUMMARY:
This study aims to evaluate the efficacy and safety of intralesional injections of candida antigen, polidocanol sclerotherapy and combined candida antigen with polidocanol in treatment of patients with common warts.

DETAILED DESCRIPTION:
Warts are benign proliferations of skin and mucosa caused by the human papillomavirus . Currently, more than 100 types of human papillomavirus have been identified, which is a non-enveloped double-stranded, circular, supercoiled DNA virus enclosed in an icosahedral capsid and comprising 72capsomers Immunotherapy in wart treatment is a type of biological therapy that uses substances to stimulate the immune system to help the body fight infected cells. This includes topical agents as imiquimod, sineacatechins, and Intralesional immunotherapy which become more preferred treatment line for several types of warts, several injectable agents have been examined such as vitamin D3, interferon alpha 2B and skin test antigens such as the candida antigen and purified protein derivatives or systemic immunotherapy as zinc, cimetidine.

Intralesional candida antigen has been successfully used in the treatment of warts with the potential advantages of promising efficacy, low cost, high safety profile, simple easy injection, association with distant response, absence of scarring and pigmentary changes and less pain than destructive therapies, and low or absent recurrence rates Treatments targeting and obliterating blood vessels such as pulsed dye laser and photodynamic therapy have been used in the treatment of common warts. Based on these observations, and the previous reports of the successful use of polidocanol in the treatment of various skin conditions with vascular components, the intralesional polidocanol therapy could be helpful in the treatment of common warts through the thrombotic occlusion and obliteration of blood vessels within the wart.

The complete and partial cure rates after intralesional polidocanol 3% injection in plantar warts were 60% and 25%, respectively

ELIGIBILITY:
Inclusion Criteria:

* Age group: >18years.
* Confirmed diagnosis by clinical and dermoscopic examination of common wart will be made.

Exclusion Criteria:

* Patients who receive any treatment for wart in the last month before the study.
* Patients with history of renal or liver disease.
* Patients with any evidence of bleeding diathesis, vaso-occulusive or thrombo-embolic disorders.
* Pregnant and lactating females.
* Patients who receive immunosuppressive therapy.
* Patients' refusal.
* Patients with history or evidenced hypersensitivity to any component used in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
size of warts | session every 2 weeks until complete clearance of warts or for a maximum of 6 treatment sessions and one month after last session
  measured by ruler) with photographic comparison at base line and before each session and one month after last session in relation to baseline lesion to detect response to therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luria L, Cardoza-Favarato G. Human Papillomavirus. 2023 Jan 16. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448132/ PMID 28846281
- [Background] Araldi RP, Sant'Ana TA, Modolo DG, de Melo TC, Spadacci-Morena DD, de Cassia Stocco R, Cerutti JM, de Souza EB. The human papillomavirus (HPV)-related cancer biology: An overview. Biomed Pharmacother. 2018 Oct;106:1537-1556. doi: 10.1016/j.biopha.2018.06.149. Epub 2018 Jul 26. PMID 30119229
- [Background] Parsi K, Exner T, Low J, Fung Ma DD, Joseph JE. In vitro effects of detergent sclerosants on clot formation and fibrinolysis. Eur J Vasc Endovasc Surg. 2011 Feb;41(2):267-77. doi: 10.1016/j.ejvs.2010.10.004. Epub 2010 Dec 22. PMID 21183368
- [Background] Hekmatjah J, Farshchian M, Grant-Kels JM, Mehregan D. The status of treatment for plantar warts in 2021: No definitive advancements in decades for a common dermatology disease. Clin Dermatol. 2021 Jul-Aug;39(4):688-694. doi: 10.1016/j.clindermatol.2021.05.024. Epub 2021 May 19. PMID 34809773